CLINICAL TRIAL: NCT05595226
Title: Effect of RT3D-TEE-guided Mitral Valve Repair on Outcomes in Patients With Degenerative Mitral Valve Disease
Acronym: TEEMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheng Liu (Other)
Responsible Party: Sponsor-Investigator, Sheng Liu, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEE-MVR Project
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Degenerative Mitral Valve Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT3D-TEE-guided mitral valve repair (Experimental): Two experienced surgeons and two experienced echocardiography technicians jointly formulated the plan for the TEE-guided mitral valve repair.
  Interventions: Procedure: RT3D-TEE-guided mitral valve repair
- Control (No Intervention)

INTERVENTIONS:
Procedure: RT3D-TEE-guided mitral valve repair — RT3D-TEE forms a surgical plan before surgery and 3 to 4 senior doctors with more than 50 cases of mitral valve repair perform the procedure.
  Arms: RT3D-TEE-guided mitral valve repair

SUMMARY:
The aim of this randomized controlled trial to investigate the effects of Real-time 3D transesophageal echocardiography (RT3D-TEE)-guided mitral valve repair on surgical failure and 1-year reoccurrence of mitral valve regurgitation in patients with degenerative mitral value disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic primary degenerative mitral regurgitation by the preoperative echocardiogram.
* Informed consent was obtained

Exclusion Criteria:

* Re-operation of mitral regurgitation
* Concurrent surgical plan for congenital heart disease, coronary artery bypass grafting, aortic valve surgery, radiofrequency ablation of atrial fibrillation and other cardiac surgeries.
* Mitral valve replacement
* Unable to undergo TEE

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite events of mitral valve repair failure and 1-year reoccurrence of mitral regurgitation | 1 year
  mitral valve repair failure, 1-year reoccurrence of mitral regurgitation

SECONDARY OUTCOMES:
Individual occurrence of composite endpoints of mitral valve repair failure and 1-year reoccurrence of mitral regurgitation | 1 year
The incidence of secondary transfer, perioperative complications | 1 year
Intraoperative conditions including extracorporeal circulation time, aortic occlusion time | 1 year
The recurrence rate of residual mitral valve regurgitation | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided